CLINICAL TRIAL: NCT03948126
Title: Prevalence of Geophagy and Knowledge About Its Health Effects Among Native Sub-Saharan Africa, Caribbean and South America Healthy Adults Living in France
Acronym: Prevalgeophagy
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2018Ao007
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Geophagia
Keywords: geophagia
MeSH Terms: conditions — Pica

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- travel medicine: Healthy adults originating from Sub-Saharan Africa, South America and the Caribbean and attending a travel medicine and international vaccination consultation in France.
  Interventions: Other: Questionnaire about geophagia (knowledge about soil/clay consumption and knowledge of the health effects of geophagy)

INTERVENTIONS:
Other: Questionnaire about geophagia (knowledge about soil/clay consumption and knowledge of the health effects of geophagy)

SUMMARY:
Since geophagy is widespread among women from Sub-Saharan Africa, South America and the Caribbean, we aimed to determine the frequency of geophagy and the level of knowledge about its health effects among healthy adults originating from these countries and attending a travel medicine and international vaccination consultation in France.

DETAILED DESCRIPTION:
Since geophagy is widespread among women from Sub-Saharan Africa, South America and the Caribbean, we aimed to determine the frequency of geophagy and the level of knowledge about its health effects among healthy adults originating from these countries and attending a travel medicine and international vaccination consultation in France.

A cross-sectional study was performed in the consultation for travel medicine and international vaccination in Reims University Hospital, France. All adult travellers who were natives of Sub Saharan Africa, South America and the Caribbean or born in France of parents from these countries were eligible to complete a confidential questionnaire about geophagy, which was defined as eating soil or clay. Descriptive analysis was performed.

ELIGIBILITY:
inclusion criteria : All adult travellers who were natives of Sub Saharan Africa, South America and the Caribbean or born in France of parents from these countries

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy adults originating from Sub-Saharan Africa, South America and the Caribbean and attending a travel medicine and international vaccination consultation in France.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of geophagia | Day 0
  percentage of adults with geophagia

SECONDARY OUTCOMES:
Awareness about iron-deficient anaemia | Day 0
  percentage of awareness about iron-deficient anaemia
Awareness about soil-transmitted intestinal parasitic infections | Day 0
  percentage of awareness about soil-transmitted intestinal parasitic infections
Awareness about constipation | Day 0
  percentage of awareness about constipation
Awareness about intestinal occlusion | Day 0
  percentage of awareness about intestinal occlusion

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Decaudin P, Kanagaratnam L, Kmiec I, Nguyen Y, Migault C, Lebrun D, Hentzien M, Bertin E, Drame M, Bani-Sadr F. Prevalence of geophagy and knowledge about its health effects among native Sub-Saharan Africa, Caribbean and South America healthy adults living in France. Eat Weight Disord. 2020 Apr;25(2):465-469. doi: 10.1007/s40519-018-0624-9. Epub 2018 Dec 13. PMID 30547293